CLINICAL TRIAL: NCT05272358
Title: Economic Evaluation of Early Management of Sarcoma Patients by the Sarcoma Reference Network (NETSARC), Exploration of Organisational and Financial Constraints
Brief Title: Economic Evaluation of Sarcoma Patients Management in France
Acronym: OPTISARC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Collaborators: Saint Etienne School of Mine (Other); Rennes University Hospital (Other); Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: OPTISARC
Record Dates: First submitted 2021-09-09; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Sarcoma
Keywords: cost effectiveness; network; organization; payment model; sarcoma; patient' management; initial surgery; multi disciplinary tumor board
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- strategy 1: sarcoma MDTB before surgery and initial management in the NETSARC network: Patients who had a sarcoma-specialized multidisciplinary tumour board (MDTB) before the initial surgery and complete initial management (including surgery) in the network (also including patients who had a sarcoma-specialized MDTB after the initial surgery and complete initial management in the network) (strategy 1)
  Interventions: Other: NETSARC network
- strategy 2: sarcoma MDTB before surgery and initial management outside the NETSARC network: Patients who had a sarcoma-specialized MDTB before the initial surgery and initial management (including surgery) outside the network (strategy 2)
  Interventions: Other: NETSARC network
- strategy 3: sarcoma MDTB after surgery and initial management outside the NETSARC network: Patients who had initial management (including surgery) outside the network and a sarcoma-specialized MDTB after initial surgery (strategy 3)
  Interventions: Other: NETSARC network
- strategy 4: No sarcoma MDTB and initial management outside the NETSARC network: Patients who had an initial management (including surgery) outside the network, without sarcoma-specialized MDTB neither before nor after the initial surgery (strategy 4).

INTERVENTIONS:
Other: NETSARC network — MDTB and/or surgery in NETSARC network
  Groups: strategy 1: sarcoma MDTB before surgery and initial management in the NETSARC network; strategy 2: sarcoma MDTB before surgery and initial management outside the NETSARC network; strategy 3: sarcoma MDTB after surgery and initial management outside the NETSARC network

SUMMARY:
The aim of this project is to (1) evaluate the efficiency of early management of sarcoma patients by the sarcoma referral network (NETSARC) vs. outside the network; (2) measure the budgetary impact of the generalization of the most cost-effective strategy across the country; (3) identify the organizational and financial constraints likely to hinder the generalization of the most cost-effective strategy and propose solutions, and finally (4) analyse the budgetary impact of a generalization of sarcoma patient care by the reference network by integrating the organizational and financial solutions proposed.

The study relies on an exhaustive national cohort of all sarcoma patients who underwent primary tumor surgery for the year 2013. Patients will be allocated to four distinct strategies, each representing a different management of sarcoma patients who had a sarcoma-specialized multidisciplinary tumor board (MDTB) before the initial surgery and complete initial management in the network (strategy 1); patients who had a sarcoma-specialized MDTB before the initial surgery and initial management outside the network (strategy 2); patients who had a sarcoma-specialized MDTB after initial surgery and initial management outside the network (strategy 3); patients who had an initial management outside the network, without sarcoma-specialized MDTB neither before nor after the initial surgery (strategy 4).

Matching of the National Health Data System (SNDS) and the NETSARC databases made it possible to include 2431 patients in the study. These databases will allow to obtain information on patients, estimate overall survival and identify healthcare consumption, which will be useful in achieving study's objectives.

DETAILED DESCRIPTION:
Introduction

Sarcomas are a large family of rare and heterogeneous tumors. As a consequence, their diagnosis and management are difficult and complex, which can lead to misdiagnosis and suboptimal patient management. Thus, in 2009, the National Cancer Institute (INCa) and the "Direction Générale de l'Offre de Soins" (DGOS) supported the creation of a sarcoma reference network (NETSARC) with the aim to guarantee optimal care for sarcoma patients. Numerous studies show that initial patients' management in the sarcoma referral network reduces the risk of death and relapse. However, the proportion of sarcoma patients initially managed within the referral network is still too low today. The aim of this project is to (1) evaluate the efficiency of early management of sarcoma patients by the sarcoma referral network vs. outside the network; (2) measure the budgetary impact of the generalization of the most cost-effective strategy across the country; (3) identify the organizational and financial constraints likely to hinder the generalization of the most cost-effective strategy and propose solutions, and finally (4) analyses the budgetary impact of a generalization of sarcoma patient care by the reference network by integrating the organizational and financial solutions proposed.

Methods and analysis

The study relies on an exhaustive national cohort of all sarcoma patients (ICD code 10 C49, C48 or C40-41) who underwent primary tumor surgery for the year 2013. Patients will be allocated to four distinct strategies, each representing a different management of sarcoma patients: patients who had a sarcoma-specialized multidisciplinary tumor board (MDTB) before the initial surgery and complete initial management in the network (strategy 1); patients who had a sarcoma-specialized MDTB before the initial surgery and initial management outside the network (strategy 2); patients who had a sarcoma-specialized MDTB after initial surgery and initial management outside the network (strategy 3); patients who had an initial management outside the network, without sarcoma-specialized MDTB neither before nor after the initial surgery (strategy 4).

Matching of the National Health Data System (SNDS) and the NETSARC databases made it possible to include 2431 patients in the study. These databases will allow to obtain information on patients, estimate overall survival and identify healthcare consumption, which will be useful to achieve study's objectives.

The evaluation of early management of operable sarcoma patients by the sarcoma reference network vs. outside the network will be based on three approaches which are both distinct and complementary in terms of decision support. (1) Firstly, an efficiency assessment based on a cost-effectiveness analysis (CEA) and a cost-utility analysis (CUA) will be carried out. The short-term CEA will use the Incremental Cost-Effectiveness Ratio (ICER) expressed as cost per life year gained, while the long-term CUA will use the ICER expressed as cost per quality-adjusted life year (QALY) gained. The efficiency analysis will be complemented by a Budget Impact Analysis (BIA) based on an estimate of the additional and avoided costs induced by the generalization of the most cost-effective strategy determined in the previous steps. (2) Next, an organizational evaluation focusing on a flow analysis will be carried out. (3) Finally, an innovative financing model will be developed to encourage inter-center cooperation.

Ethics and dissemination

The OPTISARC project will be conducted in accordance with the ethical principles of the latest version of the Declaration of Helsinki developed by the World Medical Association (WMA). This study falls within the framework of research not involving the human person, study or health assessment (RNIPH) and will be conducted in accordance with the French and European laws and regulations in force, as well as any other applicable guidelines.

This Project has obtained a favorable opinion from the "Comité d'Expertise pour les Recherches, les Etudes et les Evaluations dans le domaine de la Santé" (CEREES) and an authorization from the "Comité National Informatique et Liberté" (CNIL) allowing the access to SNDS data (DCIR and PMSI) from 2013 to 2018.

ELIGIBILITY:
Inclusion Criteria:

* Sarcoma diagnosis between 01/01/2013 and 31/12/2013
* International Classification of Diseases (ICD) code 10: C49 Malignant neoplasm of other connective and soft tissue, or C48 Malignant neoplasm of retroperitoneum and peritoneum, or C40-41 Malignant neoplasm of bone and articular cartilage of limbs)
* Surgery of the primary tumour.

Exclusion Criteria:

* Gastro intestinal stromal tumour
* Diagnosis not confirmed by the a second histological review

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of sarcoma patient diagnosed in 2013 with a surgery of initial tumour.
Sampling Method: Non-Probability Sample
Enrollment: 2431 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2024-02-08 (Estimated)

PRIMARY OUTCOMES:
Short-term cost-effectiveness analysis | 5 years
  The main objective of this study is to evaluate the short-term effectiveness (over a 5-year period) of sarcoma patient management by the sarcoma referral network vs. outside the network. A cost-effectiveness analysis (CEA) based on the Incremental Cost-Effectiveness Ratio (ICER) will be used to compare strategies 1, 2, 3 and 4.

SECONDARY OUTCOMES:
Long-term cost-utility analysis and cost-effectiveness analysis | 15 years
  In accordance with the High Authority of Health (Haute Autorité de Santé - HAS, in French) requirements, the short-term cost-effectiveness analysis (CEA) will be supplemented by a whole-life cost-utility analysis (CUA) (and a whole-life CEA) to assess the efficiency of sarcoma patient management by the sarcoma referral network vs. outside the network. More specifically, an extrapolation to a time frame of 15 years will be used to achieve this whole-life CUA. In the same way as the short-term CEA, the whole-life CUA and CEA will use the ICER to compare strategies 1, 2, 3 and 4 with each other.
Budget Impact Analysis | 5 years
  The decision to include a Budget Impact Analysis (BIA) in this study is in line with the framework agreement signed in January 2016 between the Economic Committee for Medicinal Products (Comité Economique des Produits de Santé - CEPS, in French) and the Pharmaceutical Industry (Les Entreprises du Médicament - LEEM, in French), which advises the implementation of a BIA in addition to the medico-economic study. The BIA will strictly comply with the HAS requirements presented in its methodological guide for BIA.
Organizational Assessment | 5 years
  A quantitative comparison of the pathway models of the four strategies with reference pathway models (calculation of the distance between the models) will be accomplish.
Define the incentive mechanisms most likely to neutralize the main obstacles identified in a theoretical model of cooperation | 5 years
  Measurement tool: discrete choice questionnaire (validated by an ethical committee) with several scenarios, administered to a panel of health professionals from the sarcoma expert centers and local centers.
  The objective is to reveal the preferences of professionals for different modalities of cooperation in order to maximise their willingness to modify their current practices, whether they are in reference or peripheral centres, in the direction of greater complementarity. The method used for this investigation will be based on the design, implementation and analysis of data from a discrete choice experiment. More precisely, it is a method based on stated preferences in which the respondents are placed in a hypothetical choice situation.
Pricing model | 5 years
  Measurement: in euros 2022 - Cost impact of a transition from diagnosis related groups (DRG) to bundle payment
  To establish a pricing model that can be implemented in France, to improve the quality of care by encouraging health establishments to cooperate.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Blay, PU-PH, Principal Investigator — Centre Leon Berard
Locations (25):
- France (25):
  - CHU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - CHU Saint-Pierre, La Réunion
  - Centre Oscar Lambret, Lille
  - CHU Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - CHU Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Institut de cancérologie de Lorraine, Nancy
  - Institut de Cancérologie de l'Ouest, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Cochin, Paris
  - CHU Saint-Louis, Paris
  - Institut Curie, Paris
  - Institut jean Godinot, Reims
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de Cancérologie CHU Hautepierre, Strasbourg
  - IUCT Institut Claudius Régaud, Toulouse
  - CHU Trousseau, Tours
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
No sharing of individual data